CLINICAL TRIAL: NCT06971380
Title: A Phase 2 Trial to Study Efficacy and Safety of HBI0101 (NXC-201) CART in Subjects With Multiple Myeloma and Light-Chain Amyloidosis.
Brief Title: Study of HBI0101 (NXC-201) CAR-T Therapy in Multiple Myeloma and Light-Chain Amyloidosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Polina Stepensky (Other)
Responsible Party: Sponsor-Investigator, Polina Stepensky, Prof. Polina Stepensky, Director Department of Bone Marrow Transplantation and Cancer Immunotherapy, Hadassah Medical Organization, Hadassah Medical Organization
Organization: Hadassah Medical Organization (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBI0101-02
Record Dates: First submitted 2025-04-23; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma, Refractory to Standard Treatment; Multiple Myeloma, Relapsed; Light Chain Amyloidosis
Keywords: Relapsed/Refractory Multiple Myeloma; Light-Chain Amyloidosis; B-cell maturation antigen (BCMA); Autologous CAR-T
MeSH Terms: conditions — Multiple Myeloma; Recurrence; Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CART BCMA (Experimental): Each subject subjects will receive a single dose of 800-1200 (±20%) x 10^6 HBI0101 CART cells
  Interventions: Biological: HBI0101 CART

INTERVENTIONS:
Biological: HBI0101 CART — HBI0101 CART is defined as autologous T cells transduced ex-vivo with anti-BCMA CAR retroviral vector encoding the chimeric antigen receptor (CAR) targeted to human BCMA. The HBI0101 CART may be provided fresh or cryopreserved.

SUMMARY:
A Phase II study of HBI0101 (NXC-201) BCMA-CART in Multiple Myeloma and Light-chain Amyloidosis Patients. The goal of the study is to evaluate the efficacy and safety of HBI0101 CART.

DETAILED DESCRIPTION:
Up to 180 subjects with relapsed/refractory (R/R) multiple myeloma (MM) or light chain amyloidosis (AL) will be enrolled in a single-arm, open-label, single-site Phase 2 study. Eligible subjects will undergo leukapheresis procedure to provide starting material for manufacturing of HBI0101 CART investigational product. Each eligible subject will receive a single dose of HBI0101 CART cells. Prior to administration of HBI0101 CART, the study subjects will undergo lymphodepletion. Following administration of HBI0101 CART the subjects will be hospitalized for several days and then will return for routine follow-up periodical visits until 24 months after infusion.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age at the time of signing informed consent.
2. Voluntarily signed informed consent form.
3. Diagnosis of multiple myeloma and/or light-chain amyloidosis with relapsed or refractory disease, with measurable disease at screening visit
4. Subject suffering from multiple myeloma must have been exposed to at least two prior lines of therapy including proteasome inhibitor, immunomodulatory (IMiDs) therapy or anti-CD38 antibody, or functionally high-risk patients (i.e. first relapse within 18 months of treatment initiation) may be included.

   Subject with amyloidosis must have been exposed to at least one prior line of therapy which includes proteasome inhibitor or anti-CD38 antibody, or subjects with insufficient response (i.e. not achieving a VGPR or CR after exposure to at least an anti-CD38 antibody and a proteasome inhibitor) may be included.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2.
6. Women of child-bearing potential (WCBP), defined as a sexually mature woman who has not undergone a hysterectomy or tubal ligation or who has not been naturally postmenopausal for at least 24 consecutive months, must have a negative serum pregnancy test prior to treatment. All sexually active WCBP and all sexually active male subjects must agree to use effective methods of birth control throughout the study.
7. Recovery to ≤ Grade 2 or baseline of any non-hematologic toxicities due to prior treatments, excluding alopecia and Grade 3 neuropathy.
8. Ability and willingness to adhere to the study visit schedule and all protocol requirements.
9. Subjects with relapsed multiple myeloma who have previously undergone allogenic stem cell transplantation must have no evidence of graft versus host disease after cessation of any immunosuppressive therapy for at least one month before recruitment to the study.

Exclusion Criteria:

1. Contraindication to a study treatment/procedure or is anticipated to receive treatment/procedure that may preclude performance of study procedures.
2. Known bulky central nervous system disease.
3. Inadequate hepatic function defined by aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 2.5 x upper limit of normal (ULN) and direct bilirubin > 4x ULN.
4. Inadequate renal function defined by serum creatinine clearance/estimated clearance of <20(ml/min).
5. International ratio (INR) or partial thromboplastin time (PTT) > 2 x ULN, unless on a stable dose of anticoagulant for a thromboembolic event (provided this event is not an exclusion criteria).
6. Inadequate bone marrow function defined by absolute neutrophil count (ANC) < 1000 cells/mm^3, platelet count < 30,000 mm^3, or hemoglobin < 8 g/dL. Subjects with absolute lymphocyte count < 300 cells/mm^3 may be excluded (due to potential challenges with producing CART cells), per investigator judgement.
7. Echocardiogram with left ventricular ejection fraction < 40%.
8. Ongoing treatment with chronic immunosuppressant such as cyclosporine or systemic steroids (physiological replacement doses of steroids are allowed up to 12 mg/m^2/d hydrocortisone or equivalent)
9. Significant co-morbid condition or disease which in the judgment of the Investigator would place the subject at undue risk or interfere with the study; examples include, but are not limited to, cirrhotic liver disease, sepsis, recent significant traumatic injury, and other conditions.
10. Known human immunodeficiency virus (HIV) positive status.
11. Active Hepatitis B or Hepatitis C active infection.
12. Active CMV infection.
13. Known history of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or mechanical control within 3 months.
14. Chronic atrial fibrillation with uncontrolled heart rate.
15. Second primary malignancies that has required therapy in the last 2 years or is not in complete remission.
16. Subjects who have had a venous thromboembolic event (e.g., pulmonary embolism or deep vein thrombosis) requiring anticoagulation and who meet any of the following criteria:

    1. Have been on a stable dose of anticoagulation for < 1 month (except for acute line insertion induced thrombosis.)
    2. Have had a Grade 2, 3, or 4 hemorrhage in the last 30 days
    3. Are experiencing continued symptoms from their venous thromboembolic event (e.g. continued dyspnea or oxygen requirement).
17. Pregnant or lactating women.
18. Participation in another interventional clinical trial within 30 days prior to screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2028-05-15 (Estimated); Study Completion 2030-05-15 (Estimated)

PRIMARY OUTCOMES:
Clinical response to HBI0101 CART | 24 months
  Percentage of subjects who achieved partial response (PR) or better

SECONDARY OUTCOMES:
Safety of HBI0101 CART | 24 months
  Incidence of Serious Adverse Events and Adverse Events of Special Interest related to study treatment
Overall response rate | 24 months
  Overall Response Rate is defined by proportion of subjects with Partial Response or better per International Myeloma Working Group (IMWG) Criteria for MM, and Partial Response or better per Hematologic Response Criteria for AL.
Overall survival | 24 months
  Overall Survival is defined by the date of the initial infusion of HBI010 CART cells to the date of the patient's death due to any cause. If the patient is alive or the vital status is unknown, then their data will be censored at the date they were last known to be alive.
Progression-free survival | 24 months
  Progression-Free Survival is defined as the time from the date of the initial infusion of HBI0101 CART to the date of first documented disease progression, or death due to any cause, whichever occurs first. This is defined as Stable Disease (or better) per IMWG Criteria for MM, and Partial Response or better per Hematologic Response Criteria for AL.
Duration of response | 24 months
  Duration of response is defined as the first observation of partial response (for patients undergoing bridging therapy, this may be the date of the initial CAR T-cell infusion), to the time of disease progression, with deaths from causes other than progression censored.
Disease-free survival | 24 months
  Disease-Free Survival proportion of MRD evaluable subjects who are MRD negative is defined as the duration from start of complete response until the time of relapse from complete response.
  Minimal Residual Response (MRD) is defined as the absence of clonal plasma cells on bone marrow aspirate (minimum test sensitivity to detect 1 in 105 nucleated cells (10-5 threshold)).
Persistence of HBI0101 CART cells | 24 months
  Quantification of HBI0101 CART cells in the blood over time
Organ response | 24 months
  Frequency of organ response (including cardiac, renal, and hepatic responses) in subject with Light-chain Amyloidosis

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah MO, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Asherie N, Kfir-Erenfeld S, Avni B, Assayag M, Dubnikov T, Zalcman N, Lebel E, Zimran E, Shaulov A, Pick M, Cohen Y, Avivi I, Cohen C, Gatt ME, Grisariu S, Stepensky P. Development and manufacture of novel locally produced anti-BCMA CAR T cells for the treatment of relapsed/refractory multiple myeloma: results from a phase I clinical trial. Haematologica. 2023 Jul 1;108(7):1827-1839. doi: 10.3324/haematol.2022.281628. PMID 36200421
- [Background] Kfir-Erenfeld S, Asherie N, Grisariu S, Avni B, Zimran E, Assayag M, Sharon TD, Pick M, Lebel E, Shaulov A, Cohen YC, Avivi I, Cohen CJ, Stepensky P, Gatt ME. Feasibility of a Novel Academic BCMA-CART (HBI0101) for the Treatment of Relapsed and Refractory AL Amyloidosis. Clin Cancer Res. 2022 Dec 1;28(23):5156-5166. doi: 10.1158/1078-0432.CCR-22-0637. PMID 36107221